CLINICAL TRIAL: NCT01715662
Title: WiiHOME-AMPS: A Pilot Randomized Controlled Trial to Investigate the Use of a Home-based Nintendo Wii Program for Rehabilitation in Older Adults With a Unilateral Transtibial or Transfemoral Amputation
Brief Title: A Pilot RCT to Investigate the Use of a Home-based Nintendo Wii Program for Rehabilitation in Older Adults With Lower Limb Amputation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H11-01246
Record Dates: First submitted 2012-10-15; First posted 2012-10-29 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Lower Limb Amputation
Keywords: rehabilitation; lower limb amputation; unilateral transtibial amputation; unilateral transfemoral amputation; older adults; cognitive computer games; home-based training; Nintendo Wii; virtual reality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wii.n.Walk (Experimental): Subjects (n=12) in the experimental arm (Wii.n.Walk) will be trained using the Wii Fit for 40-minute sessions, 3 times a week for a period of 4 weeks. Subjects will stand on the Wii Fit balance board and interact with the games through weight shifting or using the Wii remote controller. The intervention protocol includes: 1) Yoga (static single and double leg exercises), 2) Balance games (lateral and poster/anterior weight shifting exercises in standing), 3) Aerobics (running on spot and step class), and 4) Strength training (dynamic single and double leg exercises). The sessions will start in the clinic with a group of 3 participants and will graduate to individualized in-home training starting from week 2. For the in-clinic training sessions, a trained research assistant will administer the intervention and will provide external cueing and correction of the pose if the participants use unsafe technique.
  Interventions: Device: Wii.n.Walk
- Control (Placebo Comparator): Subjects (n=12) in the control arm will play cognitive computer games using Wii Big Brain for the same frequency and duration as the Wii.n.Walk arm. The sessions will start in the clinic with a group of 3 participants and will graduate to individualized in-home training starting from week 2. For the in-clinic sessions, a research assistant will administer the intervention and will provide supervision. Wii Big Brain is a low-cost commercially available gaming software to improve cognitive function.
  Interventions: Device: Wii Big Brain

INTERVENTIONS:
Device: Wii.n.Walk — Subjects will be trained using Nintendo Wii Fit (commercial fitness gaming software) for 40-minute sessions, 3x/week for 4 weeks. The intervention will initially be conducted in the clinic with a group of 3 participants and will graduate to in-home sessions starting from week 2.
  Arms: Wii.n.Walk
Device: Wii Big Brain — Subjects in the control group will be trained using Wii Big Brain Academy Degree program which is a low-cost commercially available gaming software to improve cognitive function. The intervention will initially be conducted in the clinic with a group of 3 participants and will graduate to in-home sessions starting from week 2.
  Arms: Control

SUMMARY:
This is a pilot randomized controlled trial to assess the feasibility of a home-based Nintendo Wii Fit program (Wii.n.Walk) to improve walking capacity in older adults with a lower limb amputation. Twenty four individuals with a unilateral below-knee or above-knee amputation will be randomly allocated to Wii.n.Walk or control arm. The Wii.n.Walk arm will receive aerobics, weight-shifting, balance games and exercises using the Wii Fit gaming technology. The control arm will receive cognitive computer games and exercises using Wii Big Brain Academy Degree program. Both groups will receive the intervention for 40-minute sessions, 3x/week for 4 weeks. The interventions will be conducted in combinations of in-clinic group (n=3) training and individualized in-home training. Outcome measurements will be completed by a blinded evaluator at baseline, end of treatment, and 3 weeks after the end of treatment.

Hypothesis: Our primary hypothesis is that Wii.n.Walk is feasible. Our primary clinical hypothesis is that participants in the Wii.n.Walk intervention group will experience an improvement in walking capacity compared to the control group. The secondary clinical hypothesis is that participants in the Wii.n.Walk group will experience an improvement in balance confidence, physical activity, number of steps taken per day, walking while talking, lower limb functioning, and locomotor capabilities.

DETAILED DESCRIPTION:
Purpose: To assess the feasibility a home-based Nintendo Wii Fit program (Wii.n.Walk) in improving walking capacity in older adults with a unilateral transtibial or transfemoral amputation. This study will provide seed data and information (e.g. sample size calculation) to leverage funds for a future RCT.

Hypothesis: Our primary hypothesis is that Wii.n.Walk is feasible. Our primary clinical hypothesis is that participants in the Wii.n.Walk intervention group will experience an improvement in walking capacity compared to the control group. The secondary clinical hypothesis is that participants in the Wii.n.Walk group will experience an improvement in balance confidence, physical activity, number of steps taken per day, walking while talking, lower limb functioning, and locomotor capabilities.

Justification: Many older Canadians are living with lower limb amputation (LLA). The prevalence of LLA is projected to double by 2050 primarily due to chronic systemic dysvascular diseases that are common with aging. Prosthetic rehabilitation programs are designed to enhance mobility primarily through gait retraining. An ideal rehabilitation program optimizes balance and lower limb strength which in turn enhance walking capacity which is an important determinant of health related quality of life in adults with LLA. Providing a rehabilitation program that is motivating and engaging is challenging because improvement requires highly repetitious task performance. In 1994-97, the cost of surgery, rehabilitation and one year follow up post LLAs varied between $86,000 to $110,000 (US) depending on the level of amputation. Shrinking health care resources often make it difficult to deliver sufficient amount of therapy to achieve standard of care, and impossible to deliver more therapy. Thus, novel methods which are practical, cost-effective, and well-received by clients are needed to deliver sufficient amounts of therapy. Commercially available gaming software such as the Wii Fit by Nintendo has the potential to be a valuable intervention for older adults with LLA. Based on pilot single subject research design study we have conducted we developed Wii.n.Walk, a home oriented intervention targeted to improve walking capacity in individuals with LLA.

Objectives: The objective of this study is to assess the feasibility of Wii.n.Walk: recruitment rate, consent rate, retention, perceived benefit from the intervention, adherence, blinding, adverse events, safety, and treatment effect.

Research Method: This is a parallel, single-blind RCT. Twenty four individuals with a unilateral transtibial or transfemoral will be randomly assigned to either the Wii.n.Walk, or the Wii Big Brain (12 in each arm) using computer-generated block randomization. The randomization will be done by a statistician who will not be involved in any part the study.

Subjects (n=12) in the Wii.n.Walk arm will be trained using the Wii Fit games for 40-minute sessions, 3 times a week for a period of 4 weeks. Subjects will stand on the Wii Fit balance board and interact with the Wii games through weight shifting or using the Wii remote controller. The intervention protocol includes: 1) Yoga (static single and double leg exercises), 2) Balance games (lateral and poster/anterior weight shifting exercises in standing), 3) Aerobics (running on spot and step class), and 4) Strength training (dynamic single and double leg exercises). For the in-clinic training sessions, a trained research assistant will administer the intervention and will provide external cueing and correction of the pose if the participants use unsafe technique.

Subjects (n=12) in the control arm will be trained using Wii Big Brain program for the same frequency and duration as the Wii.n.Walk arm. A separate research assistant will administer the intervention and will provide supervision. Wii Big Brain is a low-cost commercially available gaming software to improve cognitive function.

The interventions will be conducted in combination of in-clinic group training (n=3) and in-home individualized training.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year post a unilateral transtibial or transfemoral amputation
* 50 years of age or older
* have been using a prosthesis for at least 2 hours per day for the past 6 months
* currently not participating in another formal exercise or training program.

Exclusion Criteria:

* not able to provide an informed consent form
* not able to communicate in English
* has significant medical conditions (e.g. congestive heart failure) that contraindicates participation in exercise program
* had prosthetic socket fit issues (scores <6 on the Prosthetic Socket Fit Comfort Scale).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Two Minute Walk Test | Baseline, end of treatment, 3 weeks post treatment
  The Two Minute Walk Test (2MWT) will be used to measure walking capacity. Starting from a standing position, participants will be asked to walk as far as they can in a safe manner for two minutes over an indoor 80-meter flat out course.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, end of treatment, 3 weeks post treatment
  Short Physical Performance Battery (SPPB) will be used to measure subjects' lower extremity function by scoring their ability to perform four tasks: double-leg standing balance (feet together, semi-tandem, tandem), gait speed over 4 meters, and lower extremity strength (5x chair stands). Each task is scored from 0 (poor) to 4 (excellent). A total score will be generated by adding up the scores for individual tasks.
The Physical Activity Scale for the Elderly (PASE) | Baseline, end of treatment, 3 weeks post treatment
  The Physical Activity Scale for the Eldery (PASE) is a self-report measure that captures information on the frequency, duration, and intensity of various physical activities.
Walking While Talking Test | Baseline, end of treatment, 3 weeks post treatment
  Walking While Talking Test is a test of divided attention while locomotion. Subjects will be timed walking a 40 feet course twice while: 1) reciting the letters of the alphabet (a, b, c, ...) aloud (WWT-simple), and 2) reciting the alternate letters of the alphabet (a, c, e, …) aloud (WWT-complex). Subjects will be asked to pay attention to both walking and talking. The WWT outcomes will include total time, total numbers of alternate letters correctly recited and the total errors.
Activities-specific Balance Confidence scale (ABC) | Baseline, end of treatment, 3 weeks post treatment
  The 16-item Activities-specific Balance Confidence scale (ABC) will be used to assess self-efficacy associated with confidence to perform specific tasks without losing balance. Subjects report their confidence level on a scale of 0-100%. The individual item scores are summed and divided by 16 to derive a mean overall score with higher scores indicating higher confidence.
Modus Health StepwatchTM Activity Monitor (SAM) | Baseline, end of treatment, 3 weeks post treatment
  Modus Health StepwatchTM Activity Monitor (SAM) will be mounted on the prosthetic ankle to record number of steps taken per day.
Locomotor Capabilities Index in Amputees (LCI-5) | Baseline, end of treatment, 3 weeks post treatment
  Locomotor Capabilities Index in Amputees (LCI-5) is a subjective scale designed for people with lower limb amputation. It is composed of 14 items that ask questions about subject's ability to perform different locomotor activities with their prosthesis on. Items are scored on a 5-level ordinal scale from 0 (not able) to 4 (able to accomplish the activity alone without ambulation aids). The total score ranges from 0 to 56, with higher scores indicating greater locomotor capabilities with the prosthesis and less dependence on assistance.

OTHER OUTCOMES:
Feasibility indicators | Throughout and at the end of study
  Recruitment rate, consent rate, retention, participants' perceived benefit about the intervention, adherence, subject processing, blinding, adverse event, safety and treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: William C. Miller, PhD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Holy Family Hospital, Vancouver, British Columbia
  - GF Strong, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia